CLINICAL TRIAL: NCT07228065
Title: Pharmacy-led Intervention to Increase the Adoption of Fixed-dose Single Pill Blood Pressure Lowering Medications: Hybrid Effectiveness-Implementation Trial
Brief Title: Fixed-Dose Combinations Pragmatic Randomized Implementation Trial for Blood Pressure Control
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Julie Lauffenburger, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025P002849; 2P30AG064199 (NIH)
Record Dates: First submitted 2025-11-12; First posted 2025-11-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Primary Care
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Provider nudge only (Active Comparator): Pharmacists will deliver targeted nudges to providers through clinical decision support integrated into the EHR.
  Interventions: Behavioral: Provider nudge
- Provider nudge + Patient nudge (Experimental): In addition to provider nudges (Provider nudge only arm), patients will receive pharmacist delivered nudges (e.g., text messages) 1-7 days before the visit to encourage fixed dose combination medications.
  Interventions: Behavioral: Provider nudge; Behavioral: Patient nudge
- Provider nudge + Pharmacist collaborative practice agreement (CPA) (Experimental): In addition to provider nudges (Provider nudge only arm), patients will receive pharmacist counseling and prescribing delivered via virtual encounters after the visit.
  Interventions: Behavioral: Provider nudge; Behavioral: Pharmacist Collaborative Practice Agreement (CPA)

INTERVENTIONS:
Behavioral: Provider nudge — Pharmacists will deliver targeted nudges to providers through clinical decision support integrated into the electronic health record (EHR)
Behavioral: Patient nudge — Patients will receive pharmacist-delivered nudges (e.g., text messages) 1-7 days before their visit to encourage fixed-dosed combinations
  Arms: Provider nudge + Patient nudge
Behavioral: Pharmacist Collaborative Practice Agreement (CPA) — Patients will receive pharmacist counseling and prescribing delivered via virtual encounters after their visit
  Arms: Provider nudge + Pharmacist collaborative practice agreement (CPA)

SUMMARY:
The proposed study is an effectiveness-implementation hybrid type II trial designed to evaluate the impact of provider- and patient-directed interventions on FDC use. The trial will test the effectiveness of theory-driven nudges tailored to address provider and patient barriers. All interventions will be pharmacist-driven, with pharmacists delivering information via nudges to providers and via nudges or more intensive interventions (i.e., CPA) to patients. Data to evaluate outcomes will be extracted from electronic health records.

ELIGIBILITY:
Inclusion Criteria:

* patients with documented hypertension diagnosis
* had an elevated ambulatory blood pressure reading during the baseline visit (systolic >140 mmHg or diastolic >90 mmHg
* have an upcoming scheduled visit
* have an active prescription for 1 blood pressure lowering medication with a fixed-dose combination (FDC) alternative

Exclusion Criteria:

* in nursing homes
* already on a fixed-dose combination medication
* heart or renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure | 3 months
  Data for this outcome will be extracted from electronic health records. The primary effectiveness outcome will be a change in ambulatory systolic blood pressure at 3 months. For patients who do not return within 3 months, their index visit reading will be carried forward.

SECONDARY OUTCOMES:
Patient adoption | 3 months
  Data for this outcome will be extracted from prescription fill data that is merged with electronic health records. Adoption is defined as the proportion of patients who fill their first FDC prescription within 3 months.
Provider adoption | 3 months
  Data for this outcome will be extracted from electronic health records. Adoption will be definted as the proportion of patients whose providers prescribe FDC wtihin 3 months